CLINICAL TRIAL: NCT05565742
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of LY3819469 in Adults With Elevated Lipoprotein(a)
Brief Title: A Study of LY3819469 in Participants With Elevated Lipoprotein(a) [Lp(a)]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18547; J3L-MC-EZEB (Other: Eli Lilly and Company); 2022-501426-38-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-03; First posted 2022-10-04 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Lipoprotein Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 16 mg LY3819469 (Experimental): Participants received 16 milligrams (mg) of LY3819469 on day 1 and day 180, administered as a subcutaneous (SC) injection.
  Interventions: Drug: LY3819469
- 96 mg LY3819469 (Experimental): Participants received 96 mg of LY3819469 on day 1 and day 180, administered as a SC injection.
  Interventions: Drug: LY3819469
- 400 mg LY3819469 (Experimental): Participants received 400 mg of LY3819469 on day 1 and day 180, administered as a SC injection.
  Interventions: Drug: LY3819469
- 400 mg LY3819469 + Placebo (Experimental): Participants received 400 mg of LY3819469 on day 1 and placebo on day 180, administered as a SC injection.
  Interventions: Drug: LY3819469; Drug: Placebo
- Placebo (Placebo Comparator): Participants received placebo on day 1 and day 180, administered as a SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3819469 — Administered SC
  Arms: 16 mg LY3819469; 400 mg LY3819469; 400 mg LY3819469 + Placebo; 96 mg LY3819469
Drug: Placebo — Administered SC
  Arms: 400 mg LY3819469 + Placebo; Placebo

SUMMARY:
The main purpose of this study is to determine the efficacy and safety of LY3819469 in adults with elevated lipoprotein(a). The study will lasts about 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 40 years old at the time of signing the informed consent.
* Participants with Lp(a) ≥175 nmol/L at screening, measured at the central laboratory
* Participants on the following medications according to local practice must be on a stable regimen for at least 4 weeks prior to screening and randomization and expected to remain on a stable regimen through the end of the Treatment and Assessment Period:

  * lipid-lowering drugs
  * testosterone, estrogens, anti-estrogens, progestins, selective estrogen receptor modulators, or growth hormone
  * Have a body mass index within the range 18.5 to 40 kilogram/square meter (kg/m²), inclusive.

Male and/or Female

* Males who agree to use highly effective/effective methods of contraception may participate in this trial.
* Women not of childbearing potential (WNOCBP) may participate in this trial.

Exclusion Criteria:

* Have a history or presence of an underlying disease, or surgical, physical, medical, or psychiatric condition that, in the opinion of the investigator, would potentially affect participant safety within the study or interfere with participating in or completing the study or with the interpretation of data.
* Any of the following, or other events indicating unstable medical condition in the opinion of the investigator, within 3 months of randomization:

  * major surgery
  * coronary, carotid, or peripheral arterial revascularization
  * stroke or transient ischemic attack
  * myocardial infarction or unstable angina
  * acute limb ischemia
* Have, in the 6 months prior to day 1, uncontrolled Type 1 or Type 2 diabetes.
* Have uncontrolled hypertension

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (80):
- United States (19):
  - Care Access - 801 South Power Road, Mesa, Mesa, Arizona
  - Care Access - South Pasadena, Pasadena, California
  - Care Access - Santa Clarita, Santa Clarita, California
  - Care Access - Spring Hill, Spring Hill, Florida
  - Care Access - Pebble Beach Boulevard, Tampa, Sun City, Florida
  - Care Access - Tamarac, Tamarac, Florida
  - Care Access - Tampa, Tampa, Florida
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - Care Access - Baltimore, Baltimore, Maryland
  - Care Access - Dorchester, Dorchester, Massachusetts
  - Aventiv Research Inc, Columbus, Ohio
  - Care Access - Lima, Lima, Ohio
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley, Yardley, Pennsylvania
  - Care Access - Rapid City, Rapid City, South Dakota
  - Care Access - Georgetown, Georgetown, Texas
  - Care Access - Katy, Katy, Texas
  - Virginia Heart, Falls Church, Virginia
- Argentina (11):
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Air
  - Glenny Corp. S.A., Buenos Aires, Ciudad Aut
  - Investigaciones Medicas Imoba Srl, Balvanera, Ciudad Autónoma de Buenos Aire
  - CIPREC, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Centro Modelo de Cardiología, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán, Tucumán Province
  - CEMEDIC, Buenos Aires
  - Hospital San Roque, Córdoba
  - Centro Cardiovascular Salta, Salta
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- China (4):
  - Third People's Hospital of Hainan Province, Sanya, Hainan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
- Denmark (3):
  - Sanos Clinic, Herlev, Capital Region
  - Sanos Clinic - Nordjylland, Gandrup, North Denmark
  - Sanos Clinic - Syddanmark, Vejle, Region Syddanmark
- Germany (8):
  - Kardiologische Praxis Dr. med. univ. Wolfgang Jungmair, Bad Homburg, Hesse
  - Cardioangiologisches Centrum Bethanien, Frankfurt am Main, Hesse
  - Klinikum Bielefeld Mitte, Bielefeld, North Rhine-Westphalia
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - Medizinisches Versorgungszentrum am Bahnhof Spandau, Spandau, State of Berlin
  - Kardiologische Praxen im Spreebogen, Berlin
  - Cardiologicum Hamburg, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
- Japan (9):
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Rinku General Medical Center, Izumisano, Osaka
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Miyazaki Medical Association Hospital, Miyazaki
  - AMC Nishiumeda Clinic, Osaka
- Mexico (5):
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana, Estado de Baja California
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
- Netherlands (6):
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda, North Brabant
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Saxenburgh Medisch Centrum, Hardenberg, Overijssel
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Reinier de Graaf Ziekenhuis, locatie Delft, Delft, Zuid-Holla
  - Antonius Ziekenhuis, locatie D&A Research and Genetics, Sneek
- Romania (9):
  - Sal Med Srl, Piteşti, Argeş
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest, București
  - Centrul Medical Endocrinologie si Diabet Dr. Paveliu, Bucharest, București
  - Private Practice - Dr. Mercea Corina Delia, Baia Mare, Maramureş
  - Cardiomed, Târgu Mureş, Mureș County
  - Private Practice - Dr. Cristian Podoleanu, Târgu Mureş, Mureș County
  - Centrul Medical Medicalis, Timișoara, Timiș County
  - Cardiomed Iași, Iași
- Spain (6):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [Barcelona]
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Hospital Unviersitario Virgen Nieves, Granada
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Nissen SE, Ni W, Shen X, Wang Q, Navar AM, Nicholls SJ, Wolski K, Michael L, Haupt A, Krege JH; ALPACA Trial Investigators. Lepodisiran - A Long-Duration Small Interfering RNA Targeting Lipoprotein(a). N Engl J Med. 2025 May 1;392(17):1673-1683. doi: 10.1056/NEJMoa2415818. Epub 2025 Mar 30. PMID 40162643
- [Derived] Makhmudova U, Steinhagen-Thiessen E, Volpe M, Landmesser U. Advances in nucleic acid-targeted therapies for cardiovascular disease prevention. Cardiovasc Res. 2024 Sep 2;120(10):1107-1125. doi: 10.1093/cvr/cvae136. PMID 38970537
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- See also: A Study of LY3819469 in Participants With Elevated Lipoprotein(a) [Lp(a)] — https://trials.lilly.com/en-US/trial/363038

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
Started | 36 | 74 | 69 | 72 | 69
Received at Least One Dose of Study Drug | 36 | 74 | 69 | 72 | 69
Full Analysis Set (FAS) (All randomized participants who received at least one dose of study drug and are not discontinued due to inadvertent enrollment. Participants were analyzed according to the treatment they were assigned) | 36 | 74 | 69 | 72 | 69
Efficacy Analysis Set (EAS) (All randomized participants who received at least one dose of study drug and are not discontinued due to inadvertent enrollment. Excludes data after permanent discontinuation of study drug (for analysis post-day 180 participants were analyzed according to the treatment they were assigned) or after new initiation of medications that are known to impact Lp(a) levels.) | 36 | 74 | 69 | 72 | 69
Completed | 35 | 74 | 67 | 70 | 66
Not Completed | 1 | 0 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Participant Travelled Abroad | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 16 mg LY3819469: Participants received 16 mg of LY3819469 on day 1 and day 180, administered as a SC injection.
- Total: Total of all reporting groups
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo | Total
Number analyzed (Participants) | 36 | 74 | 69 | 72 | 69 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.55) | 63.8 (9.9) | 61.4 (10.93) | 62.2 (9.65) | 63.5 (8.42) | 62.7 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 35 | 35 | 27 | 32 | 138
  Male | 27 | 39 | 34 | 45 | 37 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 10 | 17 | 2 | 44
  Not Hispanic or Latino | 28 | 66 | 59 | 55 | 67 | 275
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 2 | 0 | 5
  Asian | 3 | 13 | 13 | 8 | 10 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 0 | 7
  White | 30 | 58 | 53 | 60 | 59 | 260
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 5 | 6 | 5 | 6 | 2 | 24
  Netherlands | 2 | 11 | 9 | 7 | 7 | 36
  Romania | 3 | 3 | 2 | 4 | 1 | 13
  United States | 8 | 17 | 19 | 19 | 24 | 87
  China | 0 | 3 | 1 | 3 | 3 | 10
  Japan | 3 | 10 | 11 | 5 | 5 | 34
  Denmark | 4 | 4 | 5 | 4 | 12 | 29
  Mexico | 2 | 0 | 2 | 4 | 0 | 8
  Germany | 5 | 12 | 8 | 6 | 10 | 41
  Spain | 4 | 8 | 7 | 14 | 5 | 38
Lipoprotein(a) [Lp(a)] level [Mean (Standard Deviation); unit: Nanomole/Liter (nmol/L)] — LPa levels were assessed using Immuno turbidimetric method.
  Nanomole/Liter (nmol/L) | 267.63 (81.80) | 278.86 (79.53) | 276.66 (100.68) | 279.98 (93.50) | 266.62 (91.31) | 274.74 (89.98)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Time Averaged Lipoprotein(a) [Lp(a)] Over Days 60-180
Description: LPa levels were assessed using Immuno turbidimetric method. Percent change is calculated as: Percent Change=[(Lp(a) at Time Point-Lp(a) at Baseline)/Lp(a) at Baseline]×100 Least squares (LS) mean was determined using mixed model repeated measures (MMRM) model with log(Lp(a)) - log(Baseline) = log(Baseline) + Treatment + Time + Treatment*Time (Type III sum of squares) as post-baseline measures. Result presented is after back-transformation. Variance-Covariance structure = Unstructured. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable.
Time Frame: Baseline, Days 60 - 180
Population: Full Analysis Set. As specified in the Protocol and statistical analysis plan (SAP), for the primary analysis up to Day 180, the two LY3819469 treatment groups assigned to 400 mg (400 mg LY3819469, 400 mg LY3819469 + placebo) were pooled into one treatment group (400 mg LY3819469 pooled) because participants received the same study intervention in the first 180 days
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled): Participants received 400 mg of LY3819469 on day 1 and day 180, administered as a SC injection.
  Participants received 400 mg of LY3819469 on day 1 and placebo on day 180, administered as a SC injection.
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) | Placebo
Number analyzed (Participants) | 36 | 74 | 141 | 69
percent change | -39.0 (7.37) | -74.4 (2.16) | -93.7 (0.38) | 3.1 (8.99)
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -40.8, 95% CI 2-sided [-55.8 to -20.6], Standard Error of Mean 8.82
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -75.2, 95% CI 2-sided [-80.4 to -68.5], Standard Error of Mean 3.01
Statistical Analysis 3: Comparison: 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -93.9, 95% CI 2-sided [-95.1 to -92.5], Standard Error of Mean 0.65

2. Secondary Outcome: Percent Change From Baseline in Time Averaged Lp(a) Over Days 240-360
Description: LPa levels were assessed using Immuno turbidimetric method. LS mean was determined using MMRM model with log(Lp(a)) - log(Baseline) = log(Baseline) + Treatment + Time + Treatment*Time (Type III sum of squares) as post-baseline measures.. Result presented is after back-transformation. Variance-Covariance structure = Unstructured. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable.
Time Frame: Baseline, Days 240 - 360
Population: Efficacy Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
Number analyzed (Participants) | 36 | 74 | 69 | 72 | 69
percent change | -38.7 (7.66) | -77.4 (1.97) | -95.0 (0.45) | -76.7 (2.06) | 0.3 (9.07)
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; LS Mean difference (Final Values) = -38.9, 95% CI 2-sided [-54.9 to -17.2], Standard Error of Mean 9.43
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -77.4, 95% CI 2-sided [-82.4 to -71.1], Standard Error of Mean 2.83
Statistical Analysis 3: Comparison: 400 mg LY3819469 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -95.0, 95% CI 2-sided [-96.1 to -93.6], Standard Error of Mean 0.64
Statistical Analysis 4: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -76.8, 95% CI 2-sided [-81.9 to -70.2], Standard Error of Mean 2.94

3. Secondary Outcome: Percentage of Participants Achieving Lp(a) <125 and <75 Nanomole/Liter (Nmol/L) at Days 60, 180
Description: Percentage of Participants Achieving Lp(a) <125 and <75 Nanomole/Liter (nmol/L) at Days 60, 180 is reported.
Time Frame: Days 60, 180
Population: Efficacy Analysis Set. Overall Number of Participants Analyzed = number of participants in each group. Number Analyzed = participants with available data at specified time points.
  As specified in the protocol and SAP, for the primary analysis up to Day 180, two LY3819469 treatment groups assigned to 400 mg (400 mg LY3819469,400 mg LY3819469 + placebo) were pooled into one treatment group (400 mg LY3819469 pooled) because participants are receiving same study intervention in the first 180 days.
Measure: Number; unit: percentage of participants
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) | Placebo
Number analyzed (Participants) | 36 | 74 | 141 | 69
percentage of participants
  Lp(a) <125 nmol/L: Day 60: number analyzed (Participants) | 35 | 73 | 137 | 68
  Lp(a) <125 nmol/L: Day 60 | 37.14 | 86.30 | 97.81 | 0.00
  Lp(a) <125 nmol/L: Day 180: number analyzed (Participants) | 35 | 72 | 132 | 66
  Lp(a) <125 nmol/L: Day 180 | 14.29 | 58.33 | 90.15 | 0.00
  Lp(a) <75 nmol/L: Day 60: number analyzed (Participants) | 35 | 73 | 137 | 68
  Lp(a) <75 nmol/L: Day 60 | 14.29 | 64.38 | 96.35 | 0.00
  Lp(a) <75 nmol/L: Day 180: number analyzed (Participants) | 35 | 72 | 132 | 66
  Lp(a) <75 nmol/L: Day 180 | 8.57 | 33.33 | 81.06 | 0.00
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 60; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 112.03, 95% CI 2-sided [6.35 to 1975.13]
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 60; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2762.52, 95% CI 2-sided [142.74 to 53463.34]
Statistical Analysis 3: Comparison: 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) vs Placebo; Lp(a) <125 nmol/L: Day 60; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 50904.09, 95% CI 2-sided [1700.95 to 1523398.10]
Statistical Analysis 4: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 180; Test type: Superiority; p = 0.026, Regression, Logistic; Odds Ratio (OR) = 27.94, 95% CI 2-sided [1.48 to 527.74]
Statistical Analysis 5: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 180; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 309.36, 95% CI 2-sided [17.99 to 5320.81]
Statistical Analysis 6: Comparison: 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) vs Placebo; Lp(a) <125 nmol/L: Day 180; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3060.16, 95% CI 2-sided [166.84 to 56127.55]
Statistical Analysis 7: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 60; Test type: Superiority; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 32.91, 95% CI 2-sided [1.70 to 635.94]
Statistical Analysis 8: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 60; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 579.62, 95% CI 2-sided [31.48 to 10673.41]
Statistical Analysis 9: Comparison: 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) vs Placebo; Lp(a) <75 nmol/L: Day 60; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14659.81, 95% CI 2-sided [646.35 to 332498.98]
Statistical Analysis 10: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 180; Test type: Superiority; p = 0.071, Regression, Logistic; Odds Ratio (OR) = 15.94, 95% CI 2-sided [0.79 to 321.21]
Statistical Analysis 11: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 180; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 86.32, 95% CI 2-sided [5.07 to 1468.36]
Statistical Analysis 12: Comparison: 400 mg LY3819469 and 400 mg LY3819469 + Placebo (400 mg LY3819469 Pooled) vs Placebo; Lp(a) <75 nmol/L: Day 180; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 956.84, 95% CI 2-sided [55.75 to 16422.76]

4. Secondary Outcome: Percentage of Participants Achieving Lp(a) <125 and <75 Nanomole/Liter (Nmol/L) at Days 240, 360, and 540
Description: Percentage of Participants Achieving Lp(a) <125 and <75 Nanomole/Liter (Nmol/L) at Days 240, 360, and 540 is reported.
Time Frame: Days 240, 360, and 540
Population: Efficacy Analysis Set. Overall Number of Participants Analyzed = number of participants in each group. Number Analyzed = participants with available data at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
Number analyzed (Participants) | 36 | 74 | 69 | 72 | 69
percentage of participants
  Lp(a) <125 nmol/L: Day 240: number analyzed (Participants) | 33 | 67 | 63 | 66 | 64
  Lp(a) <125 nmol/L: Day 240 | 36.36 | 88.06 | 98.41 | 78.79 | 1.56
  Lp(a) <125 nmol/L: Day 360: number analyzed (Participants) | 33 | 68 | 63 | 64 | 64
  Lp(a) <125 nmol/L: Day 360 | 24.24 | 58.82 | 88.89 | 59.38 | 0.00
  Lp(a) <125 nmol/L: Day 540: number analyzed (Participants) | 32 | 65 | 61 | 62 | 60
  Lp(a) <125 nmol/L: Day 540 | 9.38 | 32.31 | 75.41 | 35.48 | 0.00
  Lp(a) <75 nmol/L: Day 240: number analyzed (Participants) | 33 | 67 | 63 | 66 | 64
  Lp(a) <75 nmol/L: Day 240 | 18.18 | 76.12 | 96.83 | 65.15 | 1.56
  Lp(a) <75 nmol/L: Day 360: number analyzed (Participants) | 33 | 68 | 63 | 64 | 64
  Lp(a) <75 nmol/L: Day 360 | 6.06 | 41.18 | 82.54 | 42.19 | 0.00
  Lp(a) <75 nmol/L: Day 540: number analyzed (Participants) | 32 | 65 | 61 | 62 | 60
  Lp(a) <75 nmol/L: Day 540 | 0.00 | 16.92 | 45.90 | 16.13 | 0.00
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 32.05, 95% CI 2-sided [5.36 to 191.58]
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 602.39, 95% CI 2-sided [95.36 to 3805.22]
Statistical Analysis 3: Comparison: 400 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6953.37, 95% CI 2-sided [527.56 to 91646.24]
Statistical Analysis 4: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Lp(a) <125 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 347.76, 95% CI 2-sided [57.46 to 2104.62]
Statistical Analysis 5: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 360; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 54.99, 95% CI 2-sided [2.98 to 1015.84]
Statistical Analysis 6: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 360; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 363.15, 95% CI 2-sided [20.83 to 6332.68]
Statistical Analysis 7: Comparison: 400 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 360; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2953.53, 95% CI 2-sided [150.95 to 57790.71]
Statistical Analysis 8: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Lp(a) <125 nmol/L: Day 360; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 375.16, 95% CI 2-sided [21.46 to 6571.66]
Statistical Analysis 9: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 540; Test type: Superiority; p = 0.068, Regression, Logistic; Odds Ratio (OR) = 16.43, 95% CI 2-sided [0.81 to 331.69]
Statistical Analysis 10: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 540; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 84.97, 95% CI 2-sided [4.99 to 1447.48]
Statistical Analysis 11: Comparison: 400 mg LY3819469 vs Placebo; Lp(a) <125 nmol/L: Day 540; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 594.66, 95% CI 2-sided [33.99 to 10405.09]
Statistical Analysis 12: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Lp(a) <125 nmol/L: Day 540; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 110.17, 95% CI 2-sided [6.47 to 1875.77]
Statistical Analysis 13: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 240; Test type: Superiority; p = 0.010, Regression, Logistic; Odds Ratio (OR) = 11.61, 95% CI 2-sided [1.81 to 74.29]
Statistical Analysis 14: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 233.25, 95% CI 2-sided [39.92 to 1362.79]
Statistical Analysis 15: Comparison: 400 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3087.58, 95% CI 2-sided [331.26 to 28778.10]
Statistical Analysis 16: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Lp(a) <75 nmol/L: Day 240; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 144.58, 95% CI 2-sided [25.20 to 829.42]
Statistical Analysis 17: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 360; Test type: Superiority; p = 0.125, Regression, Logistic; Odds Ratio (OR) = 11.16, 95% CI 2-sided [0.51 to 243.85]
Statistical Analysis 18: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 360; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 148.30, 95% CI 2-sided [8.64 to 2546.89]
Statistical Analysis 19: Comparison: 400 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 360; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1431.38, 95% CI 2-sided [77.76 to 26349.86]
Statistical Analysis 20: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Lp(a) <75 nmol/L: Day 360; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 147.78, 95% CI 2-sided [8.60 to 2538.95]
Statistical Analysis 21: Comparison: 16 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 540; Test type: Superiority; p = 0.733, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.04 to 104.02]
Statistical Analysis 22: Comparison: 96 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 540; Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 34.28, 95% CI 2-sided [1.98 to 594.46]
Statistical Analysis 23: Comparison: 400 mg LY3819469 vs Placebo; Lp(a) <75 nmol/L: Day 540; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 159.77, 95% CI 2-sided [9.40 to 2716.42]
Statistical Analysis 24: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Lp(a) <75 nmol/L: Day 540; Test type: Superiority; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 37.98, 95% CI 2-sided [2.19 to 659.75]

5. Secondary Outcome: Percent Change From Baseline in Lp(a)
Description: LS mean was determined using MMRM model with log(Actual Measurement/Baseline) = log (Baseline) + High Risk CV Stratum (yes/no) + Treatment + Time + Treatment*Time (Type III sum of squares) as post-baseline measures. Variance-Covariance structure (Change from Baseline) = Unstructured. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable.
Time Frame: Baseline, Days 60, 180, 240, 360, and 540
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
Number analyzed (Participants) | 36 | 74 | 69 | 72 | 69
percent change
  Baseline, Day 60: number analyzed (Participants) | 35 | 73 | 68 | 69 | 68
  Baseline, Day 60 | -46.2 (6.04) | -80.4 (1.53) | -95.4 (0.26) | -95.4 (0.26) | 2.2 (8.29)
  Baseline, Day 180: number analyzed (Participants) | 35 | 72 | 63 | 69 | 66
  Baseline, Day 180 | -30.5 (9.17) | -65.3 (3.20) | -90.5 (0.64) | -90.5 (0.64) | 2.2 (9.78)
  Baseline, Day 240: number analyzed (Participants) | 33 | 67 | 63 | 66 | 64
  Baseline, Day 240 | -47.7 (6.63) | -84.8 (1.35) | -96.8 (0.23) | -84.9 (1.09) | -0.8 (9.10)
  Baseline, Day 360: number analyzed (Participants) | 33 | 68 | 63 | 64 | 64
  Baseline, Day 360 | -30.8 (9.19) | -67.7 (2.99) | -91.1 (0.69) | -68.1 (2.46) | -0.9 (9.53)
  Baseline, Day 540: number analyzed (Participants) | 32 | 65 | 61 | 62 | 60
  Baseline, Day 540 | -18.7 (8.56) | -45.1 (4.04) | -73.8 (1.69) | -52.8 (3.04) | 1.3 (7.76)
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -47.4, 95% CI 2-sided [-59.9 to -30.9], Standard Error of Mean 7.29
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -80.9, 95% CI 2-sided [-84.7 to -76.1], Standard Error of Mean 2.16
Statistical Analysis 3: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -95.5, 95% CI 2-sided [-96.3 to -94.5], Standard Error of Mean 0.45
Statistical Analysis 4: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -95.5, 95% CI 2-sided [-96.3 to -94.5], Standard Error of Mean 0.45
Statistical Analysis 5: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.019, Mixed Models Analysis; LS Mean difference (Final Values) = -31.9, 95% CI 2-sided [-50.6 to -6.2], Standard Error of Mean 11.10
Statistical Analysis 6: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -66.0, 95% CI 2-sided [-73.8 to -55.9], Standard Error of Mean 4.52
Statistical Analysis 7: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -90.7, 95% CI 2-sided [-92.6 to -88.3], Standard Error of Mean 1.09
Statistical Analysis 8: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 180; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -90.7, 95% CI 2-sided [-92.6 to -88.3], Standard Error of Mean 1.09
Statistical Analysis 9: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -47.3, 95% CI 2-sided [-61.3 to -28.3], Standard Error of Mean 8.25
Statistical Analysis 10: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -84.7, 95% CI 2-sided [-88.1 to -80.3], Standard Error of Mean 1.95
Statistical Analysis 11: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -96.8, 95% CI 2-sided [-97.4 to -95.9], Standard Error of Mean 0.38
Statistical Analysis 12: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -84.7, 95% CI 2-sided [-87.9 to -80.8], Standard Error of Mean 1.78
Statistical Analysis 13: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p = 0.029, Mixed Models Analysis; LS Mean difference (Final Values) = -30.2, 95% CI 2-sided [-49.4 to -3.6], Standard Error of Mean 11.45
Statistical Analysis 14: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -67.4, 95% CI 2-sided [-74.9 to -57.6], Standard Error of Mean 4.35
Statistical Analysis 15: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -91.0, 95% CI 2-sided [-92.9 to -88.5], Standard Error of Mean 1.11
Statistical Analysis 16: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 360; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -67.8, 95% CI 2-sided [-74.8 to -59.0], Standard Error of Mean 3.96
Statistical Analysis 17: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.093, Mixed Models Analysis; LS Mean difference (Final Values) = -19.7, 95% CI 2-sided [-37.8 to 3.7], Standard Error of Mean 10.45
Statistical Analysis 18: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -45.8, 95% CI 2-sided [-56.0 to -33.2], Standard Error of Mean 5.76
Statistical Analysis 19: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -74.2, 95% CI 2-sided [-78.8 to -68.5], Standard Error of Mean 2.59
Statistical Analysis 20: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 540; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -53.4, 95% CI 2-sided [-61.7 to -43.3], Standard Error of Mean 4.67

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB)
Description: LS mean was determined using MMRM model with log (Actual Measurement/Baseline) = log(Baseline) + Baseline Lp(a) stratum (<275 nmol/L vs. >=275 nmol/L) + High Risk CV Stratum (yes/no) + Treatment + Time + Treatment*Time (Type III sum of squares as post-baseline measures. Variance-Covariance structure (Change from Baseline) = Unstructured. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable.
Time Frame: Baseline, Days 60, 180, 240, 360, and 540
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
Number analyzed (Participants) | 36 | 74 | 69 | 72 | 69
percent change
  Baseline, Day 60: number analyzed (Participants) | 35 | 73 | 67 | 69 | 68
  Baseline, Day 60 | -10.2 (3.07) | -11.8 (2.10) | -13.9 (1.49) | -13.9 (1.49) | 0.2 (2.47)
  Baseline, Day 180: number analyzed (Participants) | 35 | 72 | 63 | 69 | 66
  Baseline, Day 180 | -7.0 (3.49) | -9.6 (2.37) | -12.6 (1.68) | -12.6 (1.68) | 1.3 (2.78)
  Baseline, Day 240: number analyzed (Participants) | 33 | 67 | 62 | 66 | 64
  Baseline, Day 240 | -7.6 (3.24) | -13.8 (2.11) | -14.0 (1.98) | -9.0 (2.05) | 1.8 (2.58)
  Baseline, Day 360: number analyzed (Participants) | 33 | 68 | 63 | 64 | 64
  Baseline, Day 360 | -2.9 (3.56) | -8.1 (2.35) | -10.4 (2.20) | -4.6 (2.33) | 4.3 (2.77)
  Baseline, Day 540: number analyzed (Participants) | 31 | 65 | 61 | 62 | 60
  Baseline, Day 540 | 1.4 (3.55) | -0.6 (2.42) | -9.1 (2.13) | -0.9 (2.31) | 4.3 (2.64)
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p = 0.010, Mixed Models Analysis; LS Mean difference (Final Values) = -10.4, 95% CI 2-sided [-17.5 to -2.6], Standard Error of Mean 3.74
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.9, 95% CI 2-sided [-17.7 to -5.8], Standard Error of Mean 3.02
Statistical Analysis 3: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -14.1, 95% CI 2-sided [-19.0 to -8.8], Standard Error of Mean 2.59
Statistical Analysis 4: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 60; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -14.1, 95% CI 2-sided [-19.0 to -8.8], Standard Error of Mean 2.59
Statistical Analysis 5: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.068, Mixed Models Analysis; LS Mean difference (Final Values) = -8.2, 95% CI 2-sided [-16.2 to 0.6], Standard Error of Mean 4.27
Statistical Analysis 6: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.003, Mixed Models Analysis; LS Mean difference (Final Values) = -10.7, 95% CI 2-sided [-17.1 to -3.8], Standard Error of Mean 3.40
Statistical Analysis 7: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -13.7, 95% CI 2-sided [-19.3 to -7.9], Standard Error of Mean 2.89
Statistical Analysis 8: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 180; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -13.7, 95% CI 2-sided [-19.3 to -7.9], Standard Error of Mean 2.89
Statistical Analysis 9: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p = 0.026, Mixed Models Analysis; LS Mean difference (Final Values) = -9.2, 95% CI 2-sided [-16.7 to -1.2], Standard Error of Mean 3.93
Statistical Analysis 10: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.4, 95% CI 2-sided [-21.1 to -9.3], Standard Error of Mean 2.99
Statistical Analysis 11: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.5, 95% CI 2-sided [-21.0 to -9.6], Standard Error of Mean 2.90
Statistical Analysis 12: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 240; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.6, 95% CI 2-sided [-16.3 to -4.4], Standard Error of Mean 3.03
Statistical Analysis 13: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p = 0.111, Mixed Models Analysis; LS Mean difference (Final Values) = -7.0, 95% CI 2-sided [-14.9 to 1.7], Standard Error of Mean 4.21
Statistical Analysis 14: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -12.0, 95% CI 2-sided [-18.1 to -5.3], Standard Error of Mean 3.25
Statistical Analysis 15: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -14.1, 95% CI 2-sided [-20.0 to -7.8], Standard Error of Mean 3.11
Statistical Analysis 16: Comparison: 400 mg LY3819469 + Placebo vs Placebo; 400 mg LY3819469, Placebo; Test type: Superiority; p = 0.013, Mixed Models Analysis; LS Mean difference (Final Values) = -8.6, 95% CI 2-sided [-14.9 to -1.9], Standard Error of Mean 3.30
Statistical Analysis 17: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.510, Mixed Models Analysis; LS Mean difference (Final Values) = -2.8, 95% CI 2-sided [-10.7 to 5.8], Standard Error of Mean 4.20
Statistical Analysis 18: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.173, Mixed Models Analysis; LS Mean difference (Final Values) = -4.7, 95% CI 2-sided [-11.1 to 2.1], Standard Error of Mean 3.35
Statistical Analysis 19: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -12.9, 95% CI 2-sided [-18.6 to -6.8], Standard Error of Mean 3.01
Statistical Analysis 20: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.139, Mixed Models Analysis; LS Mean difference (Final Values) = -5.0, 95% CI 2-sided [-11.2 to 1.7], Standard Error of Mean 3.27

7. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (hsCRP)
Description: hsCRP is a laboratory analyte that is an indicator of inflammation. Decreases in hsCRP represent reductions in inflammation. LS mean was determined using MMRM model with log (Actual Measurement/Baseline) = log(Baseline) + Baseline Lp(a) stratum (<275 nmol/L vs. >=275 nmol/L) + High Risk CV Stratum (yes/no) + Treatment + Time + Treatment*Time (Type III sum of squares as post-baseline measures. Variance-Covariance structure (Change from Baseline) = Unstructured. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable.
Time Frame: Baseline, Days 60, 180, 240, 360, and 540
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
Number analyzed (Participants) | 36 | 74 | 69 | 72 | 69
percent change
  Baseline, Day 60: number analyzed (Participants) | 33 | 72 | 67 | 69 | 67
  Baseline, Day 60 | -15.4 (13.94) | 0.1 (11.22) | -1.9 (8.00) | -1.9 (8.00) | 2.1 (11.87)
  Baseline, Day 180: number analyzed (Participants) | 34 | 73 | 63 | 69 | 65
  Baseline, Day 180 | 10.6 (18.22) | -6.5 (10.59) | 16.2 (9.72) | 16.2 (9.72) | 10.3 (13.17)
  Baseline, Day 240: number analyzed (Participants) | 32 | 66 | 63 | 64 | 64
  Baseline, Day 240 | -3.4 (13.02) | -8.4 (8.60) | 7.3 (9.50) | -1.2 (8.67) | 9.1 (10.52)
  Baseline, Day 360: number analyzed (Participants) | 33 | 68 | 63 | 64 | 64
  Baseline, Day 360 | 43.6 (25.21) | 13.5 (13.89) | 10.4 (12.90) | 32.3 (15.36) | 10.8 (14.04)
  Baseline, Day 540: number analyzed (Participants) | 32 | 65 | 63 | 62 | 59
  Baseline, Day 540 | -7.7 (14.93) | -1.2 (11.19) | 0.9 (11.12) | 14.1 (12.65) | 0.1 (11.89)
Statistical Analysis 1: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p = 0.353, Mixed Models Analysis; LS Mean difference (Final Values) = -17.1, 95% CI 2-sided [-44.3 to 23.3], Standard Error of Mean 16.71
Statistical Analysis 2: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p = 0.902, Mixed Models Analysis; LS Mean difference (Final Values) = -2.0, 95% CI 2-sided [-28.7 to 34.7], Standard Error of Mean 15.84
Statistical Analysis 3: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 60; Test type: Superiority; p = 0.779, Mixed Models Analysis; LS Mean difference (Final Values) = -3.9, 95% CI 2-sided [-27.4 to 27.1], Standard Error of Mean 13.65
Statistical Analysis 4: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 60; Test type: Superiority; p = 0.779, Mixed Models Analysis; LS Mean difference (Final Values) = -3.9, 95% CI 2-sided [-27.4 to 27.1], Standard Error of Mean 13.65
Statistical Analysis 5: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.987, Mixed Models Analysis; LS Mean difference (Final Values) = 0.3, 95% CI 2-sided [-32.8 to 49.7], Standard Error of Mean 20.41
Statistical Analysis 6: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.316, Mixed Models Analysis; LS Mean difference (Final Values) = -15.2, 95% CI 2-sided [-38.7 to 17.2], Standard Error of Mean 13.96
Statistical Analysis 7: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.720, Mixed Models Analysis; LS Mean difference (Final Values) = 5.4, 95% CI 2-sided [-20.9 to 40.4], Standard Error of Mean 15.37
Statistical Analysis 8: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 180; Test type: Superiority; p = 0.720, Mixed Models Analysis; LS Mean difference (Final Values) = 5.4, 95% CI 2-sided [-20.9 to 40.4], Standard Error of Mean 15.37
Statistical Analysis 9: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p = 0.461, Mixed Models Analysis; LS Mean difference (Final Values) = -11.5, 95% CI 2-sided [-36.1 to 22.6], Standard Error of Mean 14.66
Statistical Analysis 10: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p = 0.194, Mixed Models Analysis; LS Mean difference (Final Values) = -16.1, 95% CI 2-sided [-35.6 to 9.4], Standard Error of Mean 11.29
Statistical Analysis 11: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 240; Test type: Superiority; p = 0.898, Mixed Models Analysis; LS Mean difference (Final Values) = -1.7, 95% CI 2-sided [-24.0 to 27.2], Standard Error of Mean 12.87
Statistical Analysis 12: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 240; Test type: Superiority; p = 0.448, Mixed Models Analysis; LS Mean difference (Final Values) = -9.4, 95% CI 2-sided [-29.9 to 17.0], Standard Error of Mean 11.81
Statistical Analysis 13: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p = 0.233, Mixed Models Analysis; LS Mean difference (Final Values) = 29.6, 95% CI 2-sided [-15.4 to 98.4], Standard Error of Mean 28.05
Statistical Analysis 14: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p = 0.891, Mixed Models Analysis; LS Mean difference (Final Values) = 2.4, 95% CI 2-sided [-27.6 to 44.9], Standard Error of Mean 18.04
Statistical Analysis 15: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 360; Test type: Superiority; p = 0.984, Mixed Models Analysis; LS Mean difference (Final Values) = -0.4, 95% CI 2-sided [-29.0 to 39.9], Standard Error of Mean 17.18
Statistical Analysis 16: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 360; Test type: Superiority; p = 0.302, Mixed Models Analysis; LS Mean difference (Final Values) = 19.4, 95% CI 2-sided [-14.8 to 67.5], Standard Error of Mean 20.52
Statistical Analysis 17: Comparison: 16 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.684, Mixed Models Analysis; LS Mean difference (Final Values) = -7.9, 95% CI 2-sided [-37.9 to 36.8], Standard Error of Mean 18.49
Statistical Analysis 18: Comparison: 96 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.933, Mixed Models Analysis; LS Mean difference (Final Values) = -1.4, 95% CI 2-sided [-28.6 to 36.3], Standard Error of Mean 16.19
Statistical Analysis 19: Comparison: 400 mg LY3819469 vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.962, Mixed Models Analysis; LS Mean difference (Final Values) = 0.8, 95% CI 2-sided [-26.7 to 38.6], Standard Error of Mean 16.33
Statistical Analysis 20: Comparison: 400 mg LY3819469 + Placebo vs Placebo; Baseline to Day 540; Test type: Superiority; p = 0.422, Mixed Models Analysis; LS Mean difference (Final Values) = 13.9, 95% CI 2-sided [-17.2 to 56.9], Standard Error of Mean 18.52

8. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY3819469
Description: AUC was computed using the population PK model. Therefore, the concentrations are simulated from time 0 to infinity to estimate AUC for each participant. The timeframe reflects the PK timepoints that were collected to develop the population PK. Although this is a multiple dose study, the plasma PK is very short, so AUC0-180days is equivalent to AUC0-infinity.
Time Frame: Day 1: 0.5 hours, 4-9 hours post-dose; Day 180: 24-36 hours post-dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo
Number analyzed (Participants) | 35 | 74 | 69 | 72
nanogram*hour per milliliter (ng*hr/mL) | 1853 (36) | 10110 (26) | 55242 (42) | 46633 (13)

ADVERSE EVENTS:
Time Frame: Baseline Up to Day 540
Description: FAS: All randomized participants who received at least one dose of study drug and are not discontinued due to inadvertent enrollment. For safety analysis FAS was used based on actual treatment received. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 16 mg LY3819469 | 96 mg LY3819469 | 400 mg LY3819469 | 400 mg LY3819469 + Placebo | Placebo
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/74 | 0/69 | 0/72 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/36 | 9/74 | 11/69 | 8/72 | 6/69
Other Adverse Events (participants affected / at risk) | 14/36 | 25/74 | 34/69 | 35/72 | 26/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 16 mg LY3819469 (N=36) | 96 mg LY3819469 (N=74) | 400 mg LY3819469 (N=69) | 400 mg LY3819469 + Placebo (N=72) | Placebo (N=69)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 (0) | 1/35 (1) | 0/35 (0) | 0/27 (0) | 0/32 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic floor dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 16 mg LY3819469 (N=36) | 96 mg LY3819469 (N=74) | 400 mg LY3819469 (N=69) | 400 mg LY3819469 + Placebo (N=72) | Placebo (N=69)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 6 (8) | 8 (9) | 6 (6) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 5 (5) | 4 (4) | 7 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 7 (9) | 2 (3) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 6 (6) | 5 (5) | 10 (10) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (8) | 3 (3) | 6 (9) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (2) | 4 (7) | 2 (2) | 3 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 6 (6) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 3 (3) | 3 (3) | 4 (5)
Ovarian cyst (Reproductive system and breast disorders) | 1/9 (1) | 0/35 (0) | 0/35 (0) | 0/27 (0) | 0/32 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT05565742/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT05565742/SAP_002.pdf